CLINICAL TRIAL: NCT01226420
Title: A Phase II, Open-Label, Multi-Center Study to Assess the Safety and Efficacy of Alefacept in Subjects With Steroid-Refractory Chronic Graft-versus-Host Disease
Brief Title: Alefacept in Subjects With Steroid-Refractory Chronic Graft-versus-Host Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Discontinuation of drug supply from Astellas.
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Astellas Pharma Inc (Industry)
Responsible Party: Principal Investigator, Corey S. Cutler, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-230
Record Dates: First submitted 2010-10-21; First posted 2010-10-22 (Estimated); Results first posted 2013-08-13 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Chronic Graft-versus-host Disease
Keywords: GVHD; Alefacept; Amevive
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — Alefacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alefacept (Experimental): Alefacept iv
  Interventions: Drug: Alefacept

INTERVENTIONS:
Drug: Alefacept — Given intravenously Days 1 and 4 of Week 1, then subcutaneously once weekly for Weeks 2-12
  Other Names: Amevive

SUMMARY:
Alefacept is a drug tht may reduce the number of T cells in circulation. This drug has been used in the treatment of psoriasis, which is a skin disorder also caused by T cells, like chronic GVHD. Information from studies in psoriasis and in other patients with GVHD suggests that this drug may help to treat chronic GVHD. Chronic GVHD is a medical condition that can develop after allogeneic stem cell transplantation. It occurs when the donor immune cells (the "graft") attack and damage organs and tissue (the "host"). It is thought that T cells, a subtype of immune cells, are responsible for the tissue damage in chronic GVHD. In this research study we are looking to see how well Alefacept works in treating chronic GVHD that has not resolved after therapy with corticosteroids.

DETAILED DESCRIPTION:
* During the first week of treatment, participants will receive 2 doses of Alefacept intravenously (Day 1 and Day 4). During weeks 2-12, Alefacept will be given subcutaneously once weekly.
* On weeks 1, 2 and every other week through Week 12 of study treatment, participants will have a physical exam, blood tests, and be asked general health and specific questions about any problems they may be having.
* Every other week, participants will be asked to complete a questionnaire about their physical symptoms, activity level and emotional well being.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosed with cGVHD according to NIH criteria
* Active cGVHD despite treatment with corticosteroids AND one additional immunosuppressive agent for at least 4 weeks, within 52 weeks of enrollment.
* Subject is a recipient of related or unrelated BMT or PBSCT
* Subject underwent transplantation at least 6 months prior to enrollment
* Subject is on stable immunosuppressive regimen for 2 weeks prior to enrollment. Adjustment of immunosuppressive medications to maintain a therapeutic level is permitted.
* Female of child bearing potential must have a negative pregnancy test prior to first dose of alefacept and must agree to practice effective contraception during the study. Men must also agree to use adequate contraception prior to study entry and for the duration of the study.
* Meets medication restriction requirements and agrees to follow medications restrictions during study.

Exclusion Criteria:

* Received donor lymphocyte infusions in the preceding 100 days
* Currently undergoing ECP
* Subject is recipient of related or unrelated UCB
* Subject has bronchiolitis obliterans, bronchiolitis obliterans with organizing pneumonia or cryptogenic organizing pneumonia as the sole manifestation of cGVHD
* Uncontrolled intercurrent active infection.
* Absolute neutrophil count < 1000/L
* AST, ALT or total bilirubin > 2x institutional upper limit of normal unless this is a manifestation of GVHD
* Recurrent or progressive malignancy at any time after HCT, as applicable for the individual malignancy
* Subject was in any clinical study within the last 30 days
* Receipt of 5 or more prior agents to treat cGVHD
* Known hypersensitivity to alefacept or any components of the study medication
* Known to be positive for human immunodeficiency virus (HIV) antibodies
* Currently enrolled in any other study for chronic GVHD treatment and receiving treatment under the study or previous participation in this study.
* Pregnant or nursing
* Concurrent illness which, in the opinion of the Investigator, may interfere with treatment or evaluation of safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corey Cutler, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Fred Hutch Cancer Research Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Alefacept: Alefacept administration (13 doses): Days 1 and 4 (subcutaneous), Weeks 1-12 (intravenous)
Period: Overall Study
Arm/Group | Alefacept
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Alefacept
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 51 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Efficacy
Description: Proportion of patients with a favorable response, defined as a complete or partial remission at week 12 as compared to baseline in subjects with steroid refractory cGVHD.
Time Frame: 2 years
Population: All enrolled subjects
Measure: Number; unit: participants
Arm/Group | Alefacept
Number analyzed (Participants) | 6
participants | 4

2. Secondary Outcome: Safety of Alefacept Infusions in Patients With Chronic GVHD.
Description: Assess the safety of alefacept in this patient population. The number of adverse events (including hematological and non-hematological safety events) will be used for safety assessment.
Time Frame: 2 years
Population: All enrolled subjects were included in the Analysis of Safety Events
Measure: Number; unit: Total adverse events
Arm/Group | Alefacept
Number analyzed (Participants) | 6
Total adverse events | 2

ADVERSE EVENTS:
Arm/Group | Alefacept
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alefacept (N=6)
Infection (otitis externa) (Infections and infestations) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No